CLINICAL TRIAL: NCT02029898
Title: Adaptation to Neonatal Life After an Anesthetic Protocol Using Remifentanil for General Anesthesia for Caesarean Section in a Context of Prematurity - REAGI Protocol
Brief Title: Remifentanil for General Anesthesia in the Context of Immaturity
Acronym: REAGI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2012/175/HP
Record Dates: First submitted 2014-01-06; First posted 2014-01-08 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cesarean Section; Anesthesia
Keywords: cesarean section; anesthesia; children
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remifentanil (Active Comparator): injectable solution, 0.5 microgramme/Kg for 30 seconds following by a continuous dose of 0.1 microgramme/kg/minute
  Interventions: Drug: Remifentanil
- Placebo (Placebo Comparator): injectable solution 0.9% for the end of surgery
  Interventions: Drug: sodium chloride 0,9%

INTERVENTIONS:
Drug: Remifentanil
  Arms: Remifentanil
Drug: sodium chloride 0,9%
  Arms: Placebo

SUMMARY:
One of the problems during general anesthesia (GA) for caesarean section is the place of opioid agents. Indeed, the literature does not provide so far a clear answer regarding the use of opioids prior to extraction of the newborn. Indeed, if the opioid administration at induction is beneficial for the mother (better control of autonomic responses to noxious stimuli), the impact on the newborn can be unfavorable in terms of adaptation to extrauterine life . This is especially true if the birth takes place in a context of prematurity and / or acute fetal distress.

The pharmacokinetics of remifentanil make it the only opioid which is consistent with a rapid sequence induction. Its short period of action avoids the manual ventilation of patients before intubation, while providing a peak of action concomitant to the nociceptive stimulation. Patients at high risk of aspiration, including pregnant women, may benefit from this type of morphine at induction. In addition, the fact that remifentanil seems to be associated with relative fetal safety in obstetrical or neonatal context legitimized the development of protocols to study maternal-fetal consequences of the use of remifentanil at induction of AG for emergency caesarean section.

While cesarean section under general anesthesia mainly concern premature newborns in France, no work has focused on the use of remifentanil for caesarean section in a context of preterm without preeclampsia.

The main hypothesis of this study is to evaluate the safety of the use of remifentanil in terms of adaptation to extrauterine life in children born prematurely by caesarean section under general anesthesia outside the context of preeclampsia.

To do this, we will compare two groups of children, one consisting of children born by cesarean section under general anesthesia with maternal remifentanil infusion, the other made up of children born by cesarean section under general anesthesia without maternal infusion of remifentanil. This study is prospective, single-center, randomized, double-blinded.

The primary endpoint is formed by the value of the Apgar score less than 7 at 5 minutes, calculated in the delivery room by the team supporting the child (midwives and pediatricians).

The secondary endpoints are formed by maternal hemodynamic parameters (SBP, DBP, MAP, HR), the rate of complications during induction (difficult intubation, aspiration), the onset of respiratory distress requiring ventilation mask in the newborn, the rate of intubation in neonates, and the rate of use of adjuvant anesthetic agents.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria of the mother:

* Patient over 18 years
* Single pregnancy with an indication for cesarean section under general anesthesia context of prematurity (<37SA)
* Patient informed and written consent for participation in this research signed
* Affiliation to social security

Inclusion criteria of the child:

Parents informed and written consent signed by the father and mother for the participation in this research by the child (unless a parent no longer has parental authority)

Exclusion Criteria:

Non-inclusion criteria of the mother:

* Vaginal Delivery
* Mother pathology requiring the use of an opioid during induction
* Severe Preeclampsia
* More than 14 weeks between the information and the inclusion
* Patient under guardianship

Non-inclusion criteria of the child:

Fetal pathology diagnosed in the prenatal period involving the prognosis of the child

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-02-02 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2018-06-22 (Actual)

PRIMARY OUTCOMES:
Apgar Score value below 7 after 5 minutes | 5 minutes afer birth
  Apgar Score value below 7 after 5 minutes calculated in the delivery room by the team supporting the child (midwives or pediatric)

SECONDARY OUTCOMES:
Maternal hemodynamic parameters (SBP, DBP, MAP, HR), | intraoperative
Rate of complications of induction (difficult intubation, inhalation) | intraoperative
Occurrence of respiratory distress requiring mask ventilation of the newborn | intraoperative
Intubation rate among newborns | intraoperative
Rate of the use of adjuvant anesthetic agents | intraoperative
Umbilical cordon blood pH | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: TOURREL Fabien, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- CHU de Rouen, Rouen, France

REFERENCES:
- [Derived] Chollat C, Tourrel F, Houivet E, Gillet R, Verspyck E, Lecointre M, Marret S, Compere V. Low-Dose Remifentanil in Preterm Cesarean Section with General Anesthesia: A Randomized Controlled Trial. Paediatr Drugs. 2024 Jan;26(1):71-81. doi: 10.1007/s40272-023-00591-w. Epub 2023 Sep 15. PMID 37713021